CLINICAL TRIAL: NCT04194645
Title: A Randomised, Single-blind, Placebo-controlled Trial to Investigate Safety, Tolerability, and Pharmacokinetics of Single Rising Oral Doses of BI 474121 Administered as Oral Solution and Tablets to Healthy Male Subjects (SRD Part), and a Randomised, Open-label, Single-dose, Three-way Cross-over Bioavailability Comparison of BI 474121 as Tablet Versus Oral Solution and Tablet With and Without Food (BA Part)
Brief Title: A Study in Healthy Men to Test How the Body Takes up and Tolerates Different Doses of BI 474121, and Whether it Makes a Difference if BI 474121 is Taken as a Tablet or a Drink.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1411-0001; 2019-002358-22 (EudraCT Number)
Record Dates: First submitted 2019-12-10; First posted 2019-12-11 (Actual); Results first posted 2024-03-26 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (15):
- SRD: Placebo matching BI 474121 oral solution (OS) (Placebo Comparator): This arm comprises all placebo treated participants of the single rising dose (SRD) part treated with an oral solution (placebo treated participants of the two lowest dose group (DG)s). Participants receiving placebo were equally distributed across dose groups. A single dose of BI 474121 matching placebo powder for oral solution was administered after an overnight fast together with 240 milliliter (mL) of water to participants who were in a standing position.
  Interventions: Drug: Placebo solution
- SRD: Placebo matching BI 474121 tablet (T) (Placebo Comparator): This arm comprises all placebo treated participants of the SRD part treated with a tablet (placebo treated participants of the five upper DGs). Participants receiving placebo were equally distributed across dose groups. A single dose of BI 474121 matching placebo tablet was administered after an overnight fast together with 240 mL of water to subjects who were in a standing position.
  Interventions: Drug: Placebo tablet
- SRD: 0.25 milligram (mg) BI 474121 - OS (Experimental): A single dose of 0.25 mg BI 474121 was solved in 0.5 mL of water and was administered after an overnight fast together with 240 mL of water to participants who were in a standing position.
  Interventions: Drug: BI 474121 oral solution
- SRD: 1 mg BI 474121 - OS (Experimental): A single dose of 1 mg BI 474121 was solved in 2mL of water and was administered after an overnight fast together with 240 mL of water to participants who were in a standing position.
  Interventions: Drug: BI 474121 oral solution
- SRD: 2.5 mg BI 474121 - T (Experimental): A single dose of 2.5 mg BI 474121 was administered as 1 uncoated 2.5 mg tablet after an overnight fast together with 240 mL of water to participants who were in a standing position.
  Interventions: Drug: BI 474121 tablet
- SRD: 5 mg BI 474121 - T (Experimental): A single dose of 5.0 mg BI 474121 was administered as 2 uncoated 2.5 mg tablets after an overnight fast together with 240 mL of water to participants who were in a standing position.
  Interventions: Drug: BI 474121 tablet
- SRD: 10 mg BI 474121 - T (Experimental): A single dose of 10.0 mg BI 474121 was administered as 1 uncoated 10.0 mg tablet after an overnight fast together with 240 mL of water to participants who were in a standing position.
  Interventions: Drug: BI 474121 tablet
- SRD: 20 mg BI 474121 - T (Experimental): A single dose of 20.0 mg BI 474121 was administered as 2 uncoated 10.0 mg tablets after an overnight fast together with 240 mL of water to participants who were in a standing position.
  Interventions: Drug: BI 474121 tablet
- SRD: 40 mg BI 474121 - T (Experimental): A single dose of 40.0 mg BI 474121 was administered as 4 uncoated 10.0 mg tablets after an overnight fast together with 240 mL of water to participants who were in a standing position.
  Interventions: Drug: BI 474121 tablet
- BA: BI 474121 10 mg as: OS fasted (Reference (R)) / T fasted (T2) / T fed (T1) (Experimental): Participants received a single dose of 10.0 mg BI 474121 in each period, in period 1 as oral solution solved in 20 mL of water with 240 mL of water after an overnight fast (Reference (R)), in period 2 as 1 uncoated tablet with 240 mL of water after an overnight fast (Test 2 (T2)) and in period 3 as 1 uncoated tablet in fed conditions after a high-fat / high-caloric breakfast with 240 mL of water (Test 1 (T1)). Between periods was a wash-out period of at least 7 days.
  Interventions: Drug: BI 474121 tablet; Drug: BI 474121 oral solution
- BA: BI 474121 10 mg as: R / T1 / T2 (Experimental): Participants received a single dose of 10.0 mg BI 474121 in each period, in period 1 as oral solution solved in 20 mL of water with 240 mL of water after an overnight fast (R), in period 2 as 1 uncoated tablet in fed conditions after a high-fat / high-caloric breakfast with 240 mL of water (T1) and in period 3 as 1 uncoated tablet with 240 mL of water after an overnight fast (T2). Between periods was a wash-out period of at least 7 days.
  Interventions: Drug: BI 474121 tablet; Drug: BI 474121 oral solution
- BA: BI 474121 10mg as: T2 / R / T1 (Experimental): Participants received a single dose of 10.0 mg BI 474121 in each period, in period 1 as 1 uncoated tablet with 240 mL of water after an overnight fast (T2), in period 2 as oral solution solved in 20 mL of water with 240 mL of water after an overnight fast (R) and in period 3 as 1 uncoated tablet in fed conditions after a high-fat / high-caloric breakfast with 240 mL of water (T1). Between periods was a wash-out period of at least 7 days.
  Interventions: Drug: BI 474121 tablet; Drug: BI 474121 oral solution
- BA: BI 474121 10mg as: T2 / T1 / R (Experimental): Participants received a single dose of 10.0 mg BI 474121 in each period, in period 1 as 1 uncoated tablet with 240 mL of water after an overnight fast (T2), in period 2 as 1 uncoated tablet in fed conditions after a high-fat / high-caloric breakfast with 240 mL of water (T1) and in period 3 as oral solution solved in 20 mL water with 240 mL of water after an overnight fast (R). Between periods was a wash-out period of at least 7 days.
  Interventions: Drug: BI 474121 tablet; Drug: BI 474121 oral solution
- BA: BI 474121 10mg: T1 / R / T2 (Experimental): Participants received a single dose of 10.0 mg BI 474121 in each period, in period 1 as 1 uncoated tablet in fed conditions after a high-fat / high-caloric breakfast with 240 mL of water (T1), in period 2 as oral solution solved in 20 mL of water with 240 mL of water after an overnight fast (R) and in period 3 as 1 uncoated tablet with 240 mL of water after an overnight fast (T2). Between periods was a wash-out period of at least 7 days.
  Interventions: Drug: BI 474121 tablet; Drug: BI 474121 oral solution
- BA: BI 474121 10mg: T1 / T2 / R (Experimental): Participants received a single dose of 10.0 mg BI 474121 in each period, in period 1 as 1 uncoated tablet in fed conditions after a high-fat / high-caloric breakfast with 240 mL of water (T1), in period 2 as 1 uncoated tablet with 240 mL of water after an overnight fast (T2) and in period 3 as oral solution solved in 20 mL of water with 240 mL of water after an overnight fast (R). Between periods was a wash-out period of at least 7 days.
  Interventions: Drug: BI 474121 tablet; Drug: BI 474121 oral solution

INTERVENTIONS:
Drug: BI 474121 tablet — BI 474121 tablet
  Arms: BA: BI 474121 10 mg as: OS fasted (Reference (R)) / T fasted (T2) / T fed (T1); BA: BI 474121 10 mg as: R / T1 / T2; BA: BI 474121 10mg as: T2 / R / T1; BA: BI 474121 10mg as: T2 / T1 / R; BA: BI 474121 10mg: T1 / R / T2; BA: BI 474121 10mg: T1 / T2 / R; SRD: 10 mg BI 474121 - T; SRD: 2.5 mg BI 474121 - T; SRD: 20 mg BI 474121 - T; SRD: 40 mg BI 474121 - T; SRD: 5 mg BI 474121 - T
Drug: Placebo tablet — Placebo tablet
  Arms: SRD: Placebo matching BI 474121 tablet (T)
Drug: BI 474121 oral solution — BI 474121 oral solution
  Arms: BA: BI 474121 10 mg as: OS fasted (Reference (R)) / T fasted (T2) / T fed (T1); BA: BI 474121 10 mg as: R / T1 / T2; BA: BI 474121 10mg as: T2 / R / T1; BA: BI 474121 10mg as: T2 / T1 / R; BA: BI 474121 10mg: T1 / R / T2; BA: BI 474121 10mg: T1 / T2 / R; SRD: 0.25 milligram (mg) BI 474121 - OS; SRD: 1 mg BI 474121 - OS
Drug: Placebo solution — Placebo solution
  Arms: SRD: Placebo matching BI 474121 oral solution (OS)

SUMMARY:
The main objectives of this trial are to investigate safety, tolerability and pharmacokinetics (PK) of BI 474121 in healthy male subjects following oral administration of single rising doses.

ELIGIBILITY:
Inclusion criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (Blood pressure (BP), Pulse rate (PR)), 12- lead Electrocardiogram (ECG), and clinical laboratory tests
* Age of 18 to 45 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent prior to admission to the study, in accordance with Good Clinical Practice (GCP) and local legislation

Exclusion criteria:

* Any finding in the medical examination (including Blood pressure (BP), Pulse rate (PR) or Electrocardiogram (ECG)) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 100 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to the trial medication or its excipients)
* Use of drugs within 30 days of planned administration of trial medication that might reasonably influence the results of the trial (including drugs that cause QT/QTc interval prolongation)
* Intake of an investigational drug in another clinical trial within 60 days of planned administration of investigational drug in the current trial, or concurrent participation in another clinical trial in which investigational drug is administered
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day)
* Inability to refrain from smoking on specified trial days
* Alcohol abuse (consumption of more than 24 g per day)
* Drug abuse or positive drug screening
* Blood donation of more than 100 mL within 30 days of planned administration of trial medication or intended blood donation during the trial
* Intention to perform excessive physical activities within one week prior to the administration of trial medication or during the trial
* Inability to comply with the dietary regimen of the trial site
* A marked baseline prolongation of QT/QTc interval (such as QTc intervals that are repeatedly greater than 450 ms or any other relevant ECG finding at screening)
* A history of additional risk factors for Torsade de Pointes (such as heart failure, hypokalaemia, or family history of Long QT Syndrome)
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because the subject is not considered able to understand and comply with study requirements, or has a condition that would not allow safe participation in the study
* Male subjects with WOCBP partner who are unwilling to use a highly effective method of birth control from time point of administration of trial medication until 30 days thereafter.

Highly effective methods of birth control are:

* Male subject is sexually abstinent
* Male subjects is vasectomised (vasectomy at least 1 year prior to enrolment), plus condom in male subject
* Use of intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
* Use of progestogen-only hormonal contraception by female partner that inhibits ovulation (only injectables or implants), plus condom in male subject
* Use of combined (estrogen and progestogen containing) hormonal contraception by female partner that prevents ovulation (oral, intravaginal or transdermal), plus condom in male subject
* Female partner is surgically sterilised (including hysterectomy)
* Female partner is postmenopausal, defined as no menses for 1 year without an alternative medical cause (in questionable cases a blood sample with FSH above 40 U/L and estradiol below 30 ng/L is confirmatory) Sperm donation is not allowed from the time point of drug administration until 30 days thereafter.

  * ALT (alanine transaminase), AST (aspartate transaminase), or serum creatinine exceed upper limit of normal range at screening, confirmed by a repeat test
  * Orthostatic hypotension during orthostatic testing at Day -3, that the investigator considers to be of clinical relevance (only applicable for Single-rising dose (SRD) part).
  * During COVID-19 pandemic: laboratory test indicative of an ongoing SARS-CoV-2 infection.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2021-03-25 (Actual); Study Completion 2021-03-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https:// www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a two part trial in healthy male subjects: A single-blind, randomized, placebo-controlled single rising dose (SRD) scheme of BI 474121 (=SRD part); An open-label, randomized, 6-sequence cross-over to assess bioavailability (BA) of BI 474121 as oral solution (fasted state), tablet (fasted state) and tablet (fed state) (=BA part).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Participants attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Participants were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Treatment Period 1 (SRD and BA Part)
Arm/Group | SRD: Placebo Matching BI 474121 Oral Solution (OS) | SRD: Placebo Matching BI 474121 Tablet (T) | SRD: 0.25 Milligram (mg) BI 474121 - OS | SRD: 1 mg BI 474121 - OS | SRD: 2.5 mg BI 474121 - T | SRD: 5 mg BI 474121 - T | SRD: 10 mg BI 474121 - T | SRD: 20 mg BI 474121 - T | SRD: 40 mg BI 474121 - T | BA: BI 474121 10 mg as: OS Fasted (Reference (R)) / T Fasted (T2) / T Fed (T1) | BA: BI 474121 10 mg as: R / T1 / T2 | BA: BI 474121 10mg as: T2 / R / T1 | BA: BI 474121 10mg as: T2 / T1 / R | BA: BI 474121 10mg: T1 / R / T2 | BA: BI 474121 10mg: T1 / T2 / R
Started | 4 | 9 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 4 (Participants participated in the SRD part only (not in the BA part).) | 9 (Participants participated in the SRD part only (not in the BA part).) | 6 (Participants participated in the SRD part only (not in the BA part).) | 6 (Participants participated in the SRD part only (not in the BA part).) | 6 (Participants participated in the SRD part only (not in the BA part).) | 6 (Participants participated in the SRD part only (not in the BA part).) | 6 (Participants participated in the SRD part only (not in the BA part).) | 5 (Participants participated in the SRD part only (not in the BA part).) | 6 (Participants participated in the SRD part only (not in the BA part).) | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Wash-out Period 1 (BA Part Only)
Arm/Group | SRD: Placebo Matching BI 474121 Oral Solution (OS) | SRD: Placebo Matching BI 474121 Tablet (T) | SRD: 0.25 Milligram (mg) BI 474121 - OS | SRD: 1 mg BI 474121 - OS | SRD: 2.5 mg BI 474121 - T | SRD: 5 mg BI 474121 - T | SRD: 10 mg BI 474121 - T | SRD: 20 mg BI 474121 - T | SRD: 40 mg BI 474121 - T | BA: BI 474121 10 mg as: OS Fasted (Reference (R)) / T Fasted (T2) / T Fed (T1) | BA: BI 474121 10 mg as: R / T1 / T2 | BA: BI 474121 10mg as: T2 / R / T1 | BA: BI 474121 10mg as: T2 / T1 / R | BA: BI 474121 10mg: T1 / R / T2 | BA: BI 474121 10mg: T1 / T2 / R
Started | 4 (Participants participated in the SRD part only (not in the BA part).) | 9 (Participants participated in the SRD part only (not in the BA part).) | 6 (Participants participated in the SRD part only (not in the BA part).) | 6 (Participants participated in the SRD part only (not in the BA part).) | 6 (Participants participated in the SRD part only (not in the BA part).) | 6 (Participants participated in the SRD part only (not in the BA part).) | 6 (Participants participated in the SRD part only (not in the BA part).) | 5 (Participants participated in the SRD part only (not in the BA part).) | 6 (Participants participated in the SRD part only (not in the BA part).) | 2 | 2 | 2 | 2 | 2 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 4 | 9 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2 (BA Part Only)
Arm/Group | SRD: Placebo Matching BI 474121 Oral Solution (OS) | SRD: Placebo Matching BI 474121 Tablet (T) | SRD: 0.25 Milligram (mg) BI 474121 - OS | SRD: 1 mg BI 474121 - OS | SRD: 2.5 mg BI 474121 - T | SRD: 5 mg BI 474121 - T | SRD: 10 mg BI 474121 - T | SRD: 20 mg BI 474121 - T | SRD: 40 mg BI 474121 - T | BA: BI 474121 10 mg as: OS Fasted (Reference (R)) / T Fasted (T2) / T Fed (T1) | BA: BI 474121 10 mg as: R / T1 / T2 | BA: BI 474121 10mg as: T2 / R / T1 | BA: BI 474121 10mg as: T2 / T1 / R | BA: BI 474121 10mg: T1 / R / T2 | BA: BI 474121 10mg: T1 / T2 / R
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Wash-out Period 2 (BA Part Only)
Arm/Group | SRD: Placebo Matching BI 474121 Oral Solution (OS) | SRD: Placebo Matching BI 474121 Tablet (T) | SRD: 0.25 Milligram (mg) BI 474121 - OS | SRD: 1 mg BI 474121 - OS | SRD: 2.5 mg BI 474121 - T | SRD: 5 mg BI 474121 - T | SRD: 10 mg BI 474121 - T | SRD: 20 mg BI 474121 - T | SRD: 40 mg BI 474121 - T | BA: BI 474121 10 mg as: OS Fasted (Reference (R)) / T Fasted (T2) / T Fed (T1) | BA: BI 474121 10 mg as: R / T1 / T2 | BA: BI 474121 10mg as: T2 / R / T1 | BA: BI 474121 10mg as: T2 / T1 / R | BA: BI 474121 10mg: T1 / R / T2 | BA: BI 474121 10mg: T1 / T2 / R
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2 | 2 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3 (BA Part Only)
Arm/Group | SRD: Placebo Matching BI 474121 Oral Solution (OS) | SRD: Placebo Matching BI 474121 Tablet (T) | SRD: 0.25 Milligram (mg) BI 474121 - OS | SRD: 1 mg BI 474121 - OS | SRD: 2.5 mg BI 474121 - T | SRD: 5 mg BI 474121 - T | SRD: 10 mg BI 474121 - T | SRD: 20 mg BI 474121 - T | SRD: 40 mg BI 474121 - T | BA: BI 474121 10 mg as: OS Fasted (Reference (R)) / T Fasted (T2) / T Fed (T1) | BA: BI 474121 10 mg as: R / T1 / T2 | BA: BI 474121 10mg as: T2 / R / T1 | BA: BI 474121 10mg as: T2 / T1 / R | BA: BI 474121 10mg: T1 / R / T2 | BA: BI 474121 10mg: T1 / T2 / R
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 2 | 2
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS) The TS included all participants who were randomized and treated with at least 1 dose of trial drug. The treatment assignment was determined based on the first treatment the participant received. The TS was used for safety analyses.
Groups:
- SRD: 0.25 Milligram (mg) BI 474121 - OS: A single dose of 0.25 mg BI 474121 was solved in 0.5 mL water and was administered after an overnight fast together with 240 mL of water to participants who were in a standing position.
- SRD: 1 mg BI 474121 - OS: A single dose of 1 mg BI 474121 was solved in 2mL water and was administered after an overnight fast together with 240 mL of water to participants who were in a standing position.
- Total: Total of all reporting groups
Arm/Group | SRD: Placebo Matching BI 474121 Oral Solution (OS) | SRD: Placebo Matching BI 474121 Tablet (T) | SRD: 0.25 Milligram (mg) BI 474121 - OS | SRD: 1 mg BI 474121 - OS | SRD: 2.5 mg BI 474121 - T | SRD: 5 mg BI 474121 - T | SRD: 10 mg BI 474121 - T | SRD: 20 mg BI 474121 - T | SRD: 40 mg BI 474121 - T | BA: BI 474121 10 mg as: OS Fasted (Reference (R)) / T Fasted (T2) / T Fed (T1) | BA: BI 474121 10 mg as: R / T1 / T2 | BA: BI 474121 10mg as: T2 / R / T1 | BA: BI 474121 10mg as: T2 / T1 / R | BA: BI 474121 10mg: T1 / R / T2 | BA: BI 474121 10mg: T1 / T2 / R | Total
Number analyzed (Participants) | 4 | 9 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 2 | 2 | 2 | 2 | 2 | 2 | 66
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.5 (6.8) | 28.9 (4.8) | 35.2 (8.2) | 35.0 (6.4) | 31.0 (6.3) | 32.0 (7.5) | 30.5 (6.9) | 35.8 (6.5) | 32.5 (5.4) | 29.0 (5.7) | 30.5 (0.7) | 34.5 (10.6) | 36.0 (12.7) | 31.0 (1.4) | 34.0 (9.9) | 32.4 (6.4)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 4 | 9 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 2 | 2 | 2 | 2 | 2 | 2 | 66
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 9 | 6 | 6 | 6 | 6 | 6 | 5 | 6 | 2 | 2 | 2 | 2 | 2 | 2 | 66
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  White | 4 | 9 | 6 | 6 | 6 | 6 | 6 | 5 | 5 | 2 | 2 | 2 | 2 | 2 | 2 | 65
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Single Rising Dose (SRD): Percentage of Subjects With Drug-related Adverse Events.
Description: For assessment of safety and tolerability of BI 474121 the percentage of participants with drug-related adverse events (AE) was calculated.
  All AEs occurring between first drug intake till 7 days after last drug intake were assigned to the randomised treatment.
Time Frame: From drug administration until 7 days after drug administration, 7 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants
Groups:
- SRD: 1 mg BI 474121 - OS: A single dose of 1 mg BI 474121 was solved in 2 mL water and was administered after an overnight fast together with 240 mL of water to participants who were in a standing position.
Arm/Group | SRD: Placebo Matching BI 474121 Oral Solution (OS) | SRD: Placebo Matching BI 474121 Tablet (T) | SRD: 0.25 Milligram (mg) BI 474121 - OS | SRD: 1 mg BI 474121 - OS | SRD: 2.5 mg BI 474121 - T | SRD: 5 mg BI 474121 - T | SRD: 10 mg BI 474121 - T | SRD: 20 mg BI 474121 - T | SRD: 40 mg BI 474121 - T
Number analyzed (Participants) | 4 | 9 | 6 | 6 | 6 | 6 | 6 | 5 | 6
Percentage of participants | 0.0 | 11.1 | 0.0 | 0.0 | 16.7 | 16.7 | 0.0 | 20.0 | 33.3

2. Primary Outcome: Bioavailability (BA): Area Under the Concentration-time Curve of BI 474121 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz).
Description: Area under the concentration-time curve of BI 474121 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) was analyzed after single dose administration of BI 474121 as: an oral solution in fasted conditions (reference treatment), an uncoated tablet in fed conditions (treatment 1) and an uncoated tablet in fasted conditions (treatment 2).
  The geometric mean and geometric coefficient of variation were calculated by noncompartmental analysis.
Time Frame: Within 3 hours (h) before drug administration and 15 minutes (min), 30min, 1h, 1h 30min, 2h, 3h, 4h, 6h, 8h, 10h, 12h, 24h, 34h, 48h, 72h, and 96h after drug administration.
Population: Pharmacokinetic parameter analysis set (PKS):
  The PKS included all participants in the TS who provided at least 1 primary or secondary pharmacokinetic (PK) endpoint that were not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a participant was included in the PKS, even if he contributed only 1 PK parameter value for 1 period to the statistical assessment. Descriptive and model-based analyses of PK parameters were based on the PKS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour times nanomole per litre
Groups:
- BA: 10 mg BI 474121 - Oral Solution - Fasted (Reference (R)): One single dose of 10 mg BI 474121 was administered as oral solution solved in 20 milliliter (mL) of water with 240 mL of water after an overnight fast.
- BA: 10 mg BI 474121 - Tablet - Fasted (Test 2 (T2)): One single dose of 10 mg BI 474121 was administered as uncoated tablet with 240 mL of water after an overnight fast.
- BA: 10 mg BI 474121 - Tablet - Fed (Test 1 (T1)): One single dose of 10 mg BI 474121 was administered as uncoated tablet in fed conditions after a high-fat / high-caloric breakfast with 240 mL of water.
Arm/Group | BA: 10 mg BI 474121 - Oral Solution - Fasted (Reference (R)) | BA: 10 mg BI 474121 - Tablet - Fasted (Test 2 (T2)) | BA: 10 mg BI 474121 - Tablet - Fed (Test 1 (T1))
Number analyzed (Participants) | 12 | 12 | 11
Hour times nanomole per litre | 1180 (42.6) | 1150 (51.0) | 1300 (37.8)
Statistical Analysis 1: Comparison: BA: 10 mg BI 474121 - Oral Solution - Fasted (Reference (R)) vs BA: 10 mg BI 474121 - Tablet - Fasted (Test 2 (T2)); No formal hypothesis was tested; Test type: Other — The statistical model used for the analysis of the endpoint was an Analysis of Variance (ANOVA ) model on the logarithmic scale. This model included effects accounting for the following sources of variation: 'sequence', 'subjects within sequences', 'period' and 'treatment'. The effect 'subjects within sequences' was considered as random, whereas the other effects were considered as fixed; ANOVA; Ratio of geometric mean (T2/R) = 97.71, 90% CI 2-sided [91.45 to 104.40] — Intra- individual coefficient of variation (gCV %) = 8.9
Statistical Analysis 2: Comparison: BA: 10 mg BI 474121 - Tablet - Fasted (Test 2 (T2)) vs BA: 10 mg BI 474121 - Tablet - Fed (Test 1 (T1)); No formal hypothesis was tested; Test type: Other — [test comment as in outcome 2, analysis 1]; ANOVA; Ratio of geometric mean (T1/T2) = 112.88, 90% CI 2-sided [98.82 to 128.94] — Intra- individual coefficient of variation (gCV %) = 16.8

3. Primary Outcome: BA: Maximum Measured Concentration of BI 474121 in Plasma (Cmax )
Description: Maximum measured concentration of of BI 474121 in plasma (Cmax).
  The geometric mean and geometric coefficient of variation were calculated by noncompartmental analysis.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole per litre
Arm/Group | BA: 10 mg BI 474121 - Oral Solution - Fasted (Reference (R)) | BA: 10 mg BI 474121 - Tablet - Fasted (Test 2 (T2)) | BA: 10 mg BI 474121 - Tablet - Fed (Test 1 (T1))
Number analyzed (Participants) | 12 | 12 | 11
Nanomole per litre | 165 (39.6) | 79.4 (39.0) | 95.3 (22.8)
Statistical Analysis 1: Comparison: BA: 10 mg BI 474121 - Oral Solution - Fasted (Reference (R)) vs BA: 10 mg BI 474121 - Tablet - Fasted (Test 2 (T2)); No formal hypothesis was tested; Test type: Other — [test comment as in outcome 2, analysis 1]; ANOVA; Ratio of geometric mean (T2/R) = 48.02, 90% CI 2-sided [41.86 to 55.09] — Intra- individual coefficient of variation (gCV %) = 18.5
Statistical Analysis 2: Comparison: BA: 10 mg BI 474121 - Tablet - Fasted (Test 2 (T2)) vs BA: 10 mg BI 474121 - Tablet - Fed (Test 1 (T1)); No formal hypothesis was tested; Test type: Other — [test comment as in outcome 2, analysis 1]; ANOVA; Ratio of geometric mean (T1/T2) = 122.80, 90% CI 2-sided [105.04 to 143.56] — Intra- individual coefficient of variation (gCV %) = 19.8

4. Secondary Outcome: SRD: Area Under the Concentration-time Curve of BI 474121 in Plasma Over the Time Interval From 0 to the Last Quantifiable Data Point (AUC0-tz).
Description: Area under the concentration-time curve of BI 474121 in plasma over the time interval from 0 to the last quantifiable data point (AUC0-tz) was analyzed after single dose administration of BI 474121.
  The geometric mean and geometric coefficient of variation were calculated by noncompartmental analysis.
Time Frame: as for outcome 2
Population: Pharmacokinetic parameter analysis set (PKS) The PKS included all participants in the TS who provided at least 1 primary or secondary pharmacokinetic (PK) endpoint that were not excluded due to a protocol deviation relevant to the evaluation of PK or due to PK non-evaluability. Thus, a participant was included in the PKS, even if he contributed only 1 PK parameter value for 1 period to the statistical assessment. Descriptive and model-based analyses of PK parameters were based on the PKS.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour times nanomole per litre
Groups:
- SRD: 0.25 Milligram (mg) BI 474121 - Oral Solution (OS): A single dose of 0.25 milligram (mg) BI 474121 was solved in 0.5 mL water and was administered after an overnight fast together with 240 milliliter (mL) of water to participants who were in a standing position.
- SRD: 2.5 mg BI 474121 - Tablet (T): A single dose of 2.5 mg BI 474121 was administered as 1 uncoated 2.5 mg tablet after an overnight fast together with 240 mL of water to participants who were in a standing position.
Arm/Group | SRD: 0.25 Milligram (mg) BI 474121 - Oral Solution (OS) | SRD: 1 mg BI 474121 - OS | SRD: 2.5 mg BI 474121 - Tablet (T) | SRD: 5 mg BI 474121 - T | SRD: 10 mg BI 474121 - T | SRD: 20 mg BI 474121 - T | SRD: 40 mg BI 474121 - T
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 6
Hour times nanomole per litre | 31.3 (17.0) | 115 (17.1) | 314 (22.9) | 599 (33.4) | 1130 (31.0) | 2410 (31.4) | 5130 (30.2)

5. Secondary Outcome: SRD: Maximum Measured Concentration of of BI 474121 in Plasma (Cmax).
Description: as for outcome 3
Time Frame: as for outcome 2
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole per litre
Groups:
- SRD: 2.5 mg BI 474121 - Tablet (T): A single dose of 2.5 mg BI 474121 was administered as 1 uncoated 2.5 mg tablet after an overnight fast together with 240 milliliter (mL) of water to participants who were in a standing position.
- SRD: 5 mg BI 474121 - T: A single dose of 5.0 mg BI 474121 was administered as 2 uncoated 2.5 mg tablets after an overnight fast together with 240 milliliter (mL) of water to participants who were in a standing position.
- SRD: 10 mg BI 474121 - T: A single dose of 10.0 mg BI 474121 was administered as 1 uncoated 10.0 mg tablet after an overnight fast together with 240 milliliter (mL) of water to participants who were in a standing position.
- SRD: 20 mg BI 474121 - T: A single dose of 20.0 mg BI 474121 was administered as 2 uncoated 10.0 mg tablets after an overnight fast together with 240 milliliter (mL) of water to participants who were in a standing position.
- SRD: 40 mg BI 474121 - T: A single dose of 40.0 mg BI 474121 was administered as 4 uncoated 10.0 mg tablets after an overnight fast together with 240 milliliter (mL) of water to participants who were in a standing position.
Arm/Group | SRD: 0.25 Milligram (mg) BI 474121 - Oral Solution (OS) | SRD: 1 mg BI 474121 - OS | SRD: 2.5 mg BI 474121 - Tablet (T) | SRD: 5 mg BI 474121 - T | SRD: 10 mg BI 474121 - T | SRD: 20 mg BI 474121 - T | SRD: 40 mg BI 474121 - T
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 5 | 6
Nanomole per litre | 5.40 (26.3) | 19.4 (16.9) | 24.8 (12.6) | 44.3 (7.19) | 77.8 (29.4) | 189 (40.0) | 298 (29.2)

6. Secondary Outcome: BA: Area Under the Concentration-time Curve of BI 474121 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞).
Description: Area under the concentration-time curve of BI 474121 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  The geometric mean and geometric coefficient of variation were calculated by noncompartmental analysis.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour times nanomole per litre
Arm/Group | BA: 10 mg BI 474121 - Oral Solution - Fasted (Reference (R)) | BA: 10 mg BI 474121 - Tablet - Fasted (Test 2 (T2)) | BA: 10 mg BI 474121 - Tablet - Fed (Test 1 (T1))
Number analyzed (Participants) | 12 | 12 | 11
Hour times nanomole per litre | 1210 (45.0) | 1190 (53.6) | 1340 (41.0)
Statistical Analysis 1: Comparison: BA: 10 mg BI 474121 - Oral Solution - Fasted (Reference (R)) vs BA: 10 mg BI 474121 - Tablet - Fasted (Test 2 (T2)); No formal hypothesis was tested; Test type: Other — [test comment as in outcome 2, analysis 1]; ANOVA; Ratio of geometric mean (T2/R) = 98.32, 90% CI 2-sided [91.98 to 105.09] — Intra- individual coefficient of variation (gCV %) = 8.9
Statistical Analysis 2: Comparison: BA: 10 mg BI 474121 - Tablet - Fasted (Test 2 (T2)) vs BA: 10 mg BI 474121 - Tablet - Fed (Test 1 (T1)); No formal hypothesis was tested; Test type: Other — [test comment as in outcome 2, analysis 1]; ANOVA; Ratio of geometric mean (T1/T2) = 112.94, 90% CI 2-sided [98.75 to 129.18] — Intra- individual coefficient of variation (gCV %) = 16.9

ADVERSE EVENTS:
Time Frame: SRD part: From drug administration until the end of residual effect period, up to 168 hours (7 days). BA part: From drug administration until the end of residual effect period, up to 168 hours (7 days).
Groups:
- SRD: Placebo Matching BI 474121 Tablet (T): This arm comprises all placebo treated participants of the single rising dose (SRD) part treated with a tablet (placebo treated participants of the five upper DGs). Participants receiving placebo were equally distributed across dose groups. A single dose of BI 474121 matching placebo tablet was administered after an overnight fast together with 240 mL of water to subjects who were in a standing position.
Arm/Group | SRD: Placebo Matching BI 474121 Oral Solution (OS) | SRD: Placebo Matching BI 474121 Tablet (T) | SRD: 0.25 Milligram (mg) BI 474121 - OS | SRD: 1 mg BI 474121 - OS | SRD: 2.5 mg BI 474121 - T | SRD: 5 mg BI 474121 - T | SRD: 10 mg BI 474121 - T | SRD: 20 mg BI 474121 - T | SRD: 40 mg BI 474121 - T | BA: 10 mg BI 474121 - Oral Solution - Fasted (Reference (R)) | BA: 10 mg BI 474121 - Tablet - Fasted (Test 2 (T2)) | BA: 10 mg BI 474121 - Tablet - Fed (Test 1 (T1))
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/9 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/12 | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/9 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6 | 0/12 | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/4 | 4/9 | 0/6 | 1/6 | 2/6 | 1/6 | 0/6 | 1/5 | 3/6 | 3/12 | 3/12 | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | SRD: Placebo Matching BI 474121 Oral Solution (OS) (N=4) | SRD: Placebo Matching BI 474121 Tablet (T) (N=9) | SRD: 0.25 Milligram (mg) BI 474121 - OS (N=6) | SRD: 1 mg BI 474121 - OS (N=6) | SRD: 2.5 mg BI 474121 - T (N=6) | SRD: 5 mg BI 474121 - T (N=6) | SRD: 10 mg BI 474121 - T (N=6) | SRD: 20 mg BI 474121 - T (N=5) | SRD: 40 mg BI 474121 - T (N=6) | BA: 10 mg BI 474121 - Oral Solution - Fasted (Reference (R)) (N=12) | BA: 10 mg BI 474121 - Tablet - Fasted (Test 2 (T2)) (N=12) | BA: 10 mg BI 474121 - Tablet - Fed (Test 1 (T1)) (N=11)
Photophobia (Eye disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 2 | 2 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Initial insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to the current COVID-19 pandemic, the recruitment of new subjects was temporarily discontinued. Ongoing, randomised patients were managed as per Trial Protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/45/NCT04194645/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/45/NCT04194645/SAP_001.pdf